CLINICAL TRIAL: NCT03552237
Title: The Effect of Dietary Fiber Supplement on the Intestinal Microbiota Among Schizophrenia Patients With Central Obesity: a Pilot Study
Brief Title: Effect of Dietary Fiber Supplement on the Intestinal Microbiota Among Schizophrenia Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: TsaoTun Psychiatric Center, Department of Health, Taiwan (Other)
Responsible Party: Principal Investigator, C Lin, Director of General Psychiatry Department, TsaoTun Psychiatric Center, Department of Health, Taiwan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 106035
Record Dates: First submitted 2018-05-15; First posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Schizophrenia; Central Obesity
MeSH Terms: conditions — Schizophrenia; Obesity, Abdominal | interventions — Dietary Fiber

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dietary fiber intervention group (Experimental)
  Interventions: Dietary Supplement: dietary fiber

INTERVENTIONS:
Dietary Supplement: dietary fiber — We will investigate in a 4 week intervention whether consumption of dietary fiber supplement affect the microbiota composition in schizophrenia patients with central obesity.

SUMMARY:
Background There has been much interest in the relationship between the types of gut microbiota and the development of obesity in recent years. It has been reported that the proportions of Firmicutes and Bacteroidetes differ between obese and normal weight human subjects. Human intestinal microbiota compositions have been found to be associated with long-term dietary habits and lifestyle. However, an increasing number of researches show that intestinal microbiota composition may be affected after short-term diet intervention. Importantly, obesity and metabolic problems play important roles in morbidity and mortality of schizophrenia patients. Human intestinal microbiota compositions related with obesity may impact the heath of this population. Therefore, we searched current advances about the connection of obesity, intestinal microbiota compositions, and diet in schizophrenia to conduct a clinical research focus on the effect of high fiber diet on the intestinal microbiota of schizophrenia patients with central obesity.

Method We will investigate in a 4-week intervention whether consumption of dietary fiber supplement(Inulin) affect the microbiota composition in schizophrenia inpatients with central obesity. Fecal samples from participants before and after the intervention will be processed for the microbiota analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Schizophrenia inpatients
2. Overweight and with central obesity
3. agree to sign informed consent

Exclusion Criteria:

1. Diagnosis of IBS
2. Systemic antibiotic use during the past 4 weeks
3. Excessive water intake

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-06-20 (Estimated); Primary Completion 2018-09-20 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in microbiota composition at week 4 | 4 weeks
  Fecal samples from participants before and after the intervention will be processed for microbiota analysis